CLINICAL TRIAL: NCT04041128
Title: Pre-Surgical Window Pilot Investigation of the Effect of PARP Inhibition on the Cellular and Molecular Changes in Primary Ovarian and Breast Cancer
Brief Title: PARP Inhibition During Pre-surgical Window in Breast/Ovary Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jayanthi Lea, PROFESSOR - Obstetrics & Gynecology - OB-Gynecologic Oncology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU-2019-0769
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer; Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lynparza (Experimental): Lynparza taken orally at a dose of 300mg twice daily for 7 days
  Interventions: Drug: Lynparza

INTERVENTIONS:
Drug: Lynparza — Lynparza taken orally at a dose of 300mg twice daily for 7 days
  Other Names: Olaparib

SUMMARY:
Study involves surgery for cytoreduction or laparoscopy to determine if you are a candidate for tumor debulking or a tissue biopsy. Following this surgery you will receive chemotherapy. This study will administer 7 days of treatment with a targeted therapy called Lynparza. Lynparza and/or other PARP inhibitors have been FDA approved for the treatment of ovarian and breast cancer. Tissue biopsy will be done before a 7 day course of Lynparza in order to correlate molecular changes to response to treatment. Participation in this trial will require an additional tumor biopsy which will occur either before or after treatment of Lynparza.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have cytology/ biopsy proven diagnosis of a mullerian carcinoma, high clinical index of suspicion for ovarian cancer OR triple negative, BRCA mutated breast cancer.
* Patients may not have received prior treatment for breast or ovarian cancer.
* All patients must be of at least 18 years of age.
* ECOG Performance status must be 0,1 or 2.
* Patients must not have received a prior PARP inhibitor
* Adequate organ and marrow function as defined below:
* absolute neutrophil count >/= 1500/mcL
* Platelets > /= 100,000 /mcl
* Hemoglobin >/= 8 g/dl
* Total bilirubin </= 1.5 x the institutional ULN
* AST, ALT </= 3 x the institutional ULN
* Creatinine </= the institutional ULN
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Patients must be able to swallow and retain oral medications.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Chemotherapy, radiotherapy, or other cancer therapy within 4 weeks prior to starting study treatment. Subjects must have recovered from prior treatment-related to toxicities to grade 1 or baseline (excluding alopecia and clinically stable toxicities requiring ongoing medical management, such as hypothyroidism from prior immune checkpoint inhibitor treatment).
* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* Brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Lynparza or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Measure DNA damage response to PARP inhibition | Following 7 days of Lynparza
  Paired t-test or Wilcoxon signed-rank test will be used to examine if there is a significant change in ADP ribosylated proteome, DNA damage, apoptosis and change in RAD 51 foci between pre-and post-treatment cancer specimens.
Characterize changes in ADP ribosylation to PARP inhibition | Following 7 days of Lynparza
  Spearman rank correlation will be computed to estimate the correlation between the changes in ADP ribosylation with the response (measured by immunohistochemistry: γH2AX and caspase -3 cleavage)
Correlate DNA damage response to ADP ribosylated proteome | Following 7 days of Lynparza
  Paired t-test or Wilcoxon signed-rank test will be used to examine if there is a significant change in ADP ribosylated proteome, DNA damage, apoptosis and change in RAD 51 foci between pre-and post-treatment cancer specimens

CONTACTS AND LOCATIONS:
Overall Officials: Jayanthi Lea, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States